CLINICAL TRIAL: NCT00825084
Title: A Phase 1, Randomized, Subject- And Investigator-Blind, Sponsor-Open, Placebo-Controlled, Parallel-Cohort, Single-Dose Escalation, And Multiple-Dose Titration Study To Evaluate The Pharmacokinetics, Safety, And Tolerability Of Dimebon [PF-01913539] In Japanese And Western Healthy Subjects
Brief Title: A Phase 1 Study To Evaluate The Pharmacokinetics, Safety, And Tolerability Of Dimebon [PF-01913539] In Japanese And Western Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1451014
Record Dates: First submitted 2009-01-12; First posted 2009-01-19 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Alzheimer's Disease; Huntington's Disease
Keywords: Dimebon, Japanese and Western population, pharmacokinetics
MeSH Terms: conditions — Alzheimer Disease; Huntington Disease | interventions — latrepirdine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- single dose cohort-Japanese group (Experimental): Japanese healthy subjects
  Interventions: Drug: Dimebon
- single dose cohort-Western group (Experimental): Western healthy subjects
  Interventions: Drug: Dimebon
- multiple dose cohort-Japanese group (Experimental): Japanese healthy subjects
  Interventions: Drug: Dimebon
- multiple dose cohort-Western group (Experimental): Western healthy subjects
  Interventions: Drug: Dimebon

INTERVENTIONS:
Drug: Dimebon — dose escalation of single oral doses of 5, 10 and 20 mg
  Arms: single dose cohort-Japanese group
Drug: Dimebon — dose escalation of single oral doses of 5, 10 and 20 mg
  Arms: single dose cohort-Western group
Drug: Dimebon — 10 mg TID of Dimebon for 7 days followed by 20 mg TID of Dimebon for 7 days
  Arms: multiple dose cohort-Japanese group
Drug: Dimebon — 10 mg TID of Dimebon for 7 days followed by 20 mg TID of Dimebon for 7 days
  Arms: multiple dose cohort-Western group

SUMMARY:
This study is to characterize the pharmacokinetics of single and multiple oral doses of Dimebon in Japanese healthy subjects. This study is also to evaluate the safety and tolerability of single and multiple oral doses of Dimebon in Japanese healthy subjects. The secondary objective of this study is to compare the pharmacokinetics, safety and tolerability of single and multiple oral doses of Dimebon in Japanese and Western healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG, and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight within the range of 50 to 100 kg.
* An informed consent document signed and dated by the subject or a legally-acceptable representative.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Japanese subjects must have four Japanese grandparents who were born in Japan.

Exclusion Criteria:

* Asian or Polynesian subjects in Western subject groups.
* Any condition possibly affecting drug absorption (e.g., gastrectomy, active peptic ulcer within last 3 months).
* History of regular alcohol consumption exceeding an average of 7 drinks/week for females and 14 drinks/week for men (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* Subjects who, by history, smoke more than 5 cigarettes per day.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
* 12-lead ECG demonstrating QTc >450 msec at screening. If QTc exceeds 450 msec, the ECG may be repeated two more times and the average of the three QTc values should be used to determine the subject's eligibility.
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of nonhormonal contraception as outlined in this protocol from at least 14 days prior to the first dose of study medication.
* Use of prescription or nonprescription drugs, vitamins and dietary supplements, within 7 days or 5 half-lives (whichever is longer) of the first dose of study medication. Herbal supplements and hormonal methods of contraception (including oral and transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone-releasing IUDs, postcoital contraceptive methods) and hormone replacement therapy must be discontinued 28 days prior to the first dose of study medication. Depo-Provera® must be discontinued at least 6 months prior to the first dose of study medication. As an exception, acetaminophen/paracetamol may be used at doses of ≤ 2 grams/day. Limited use of non-prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2009-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
plasma drug concentrations | 72 hours post last dose

SECONDARY OUTCOMES:
Safety will be including physical/neurological examination findings, clinical safety laboratory assessments, 12-lead ECGs, vital sign measurements and adverse event monitoring | 72 hours post last dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Glendale, California, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1451014&StudyName=A%20Phase%201%20Study%20To%20Evaluate%20The%20Pharmacokinetics%2C%20Safety%2C%20And%20Tolerability%20Of%20Dimebon%20%5BPF-01913539%5D%20In%20Japanese%20And%20Western%20Health